CLINICAL TRIAL: NCT00000821
Title: Subcutaneously Administered Aldesleukin ( Interleukin-2; IL-2 ) Therapy in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: IRP 015; IL-2 SC; 93-I-0205
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interleukin-2; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
To compare the effects of low-dose versus high-dose subcutaneous ( SC ) aldesleukin ( interleukin-2; IL-2 ) on immunologic and virologic markers in HIV-infected patients. To compare the effects of monthly versus bimonthly administration of SC IL-2 on these markers.

Interleukin-2 is a protein that is naturally produced by lymphocytes. In an initial study, patients in an earlier stage of HIV-1 infection tended to tolerate SC IL-2 better than those with more advanced infections, and those with higher baseline CD4+ counts tended to derive the greatest benefit.

DETAILED DESCRIPTION:
Interleukin-2 is a protein that is naturally produced by lymphocytes. In an initial study, patients in an earlier stage of HIV-1 infection tended to tolerate SC IL-2 better than those with more advanced infections, and those with higher baseline CD4+ counts tended to derive the greatest benefit.

Patients are randomized to one of four treatment arms; patients receive either low-dose or high-dose SC IL-2 for 5 days either on a monthly or bimonthly schedule for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity.
* CD4 count >= 500 cells/mm3.
* No history of AIDS-defining opportunistic infection, or malignancy other than mucocutaneous Kaposi's sarcoma.

Concurrent Medication: Required:

* Concurrent FDA-approved antiretroviral therapy (AZT, ddI, ddC, d4T).

Prior Medication: Required:

* FDA-approved antiretroviral therapy for at least 6 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant cardiac, pulmonary, thyroid, renal, or CNS disease.

Prior Medication:

Excluded:

* Prior IL-2.
* Systemic corticosteroids, chemotherapy, or experimental therapy within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Natl Inst of Allergy & Infect Dis / Cln Ctr, Bethesda, Maryland, United States

REFERENCES:
- [Background] Giedlin M, McGrath M, Gascon R, DeGroat S, Fyfe G, Kahn J. Immunological characterization of HIV seropositive patients treated with subcutaneous Proleukin (aldesleukin) recombinant Interleukin-2. Int Conf AIDS. 1996 Jul 7-12;11(2):282 (abstract no ThB4183)
- [Background] Davey RT Jr, Chaitt DG, Albert JM, Piscitelli SC, Kovacs JA, Walker RE, Falloon J, Polis MA, Metcalf JA, Masur H, Dewar R, Baseler M, Fyfe G, Giedlin MA, Lane HC. A randomized trial of high- versus low-dose subcutaneous interleukin-2 outpatient therapy for early human immunodeficiency virus type 1 infection. J Infect Dis. 1999 Apr;179(4):849-58. doi: 10.1086/314678. PMID 10068580